CLINICAL TRIAL: NCT04016623
Title: Clinical Evaluation of Invigor Toric 1-Day Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CV-19-27
Record Dates: First submitted 2019-05-14; First posted 2019-07-11 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism | interventions — Contact Lenses

STUDY DESIGN:
Intervention Model Description: This is a non-dispensing, double-masked, randomized, contralateral study design. Each subject will be randomized to wear the test lens in one eye and the control lens in the other eye.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 1-day toric test contact lens (Experimental): Each subject will wear the 1-day toric test (Test) lens in one eye and 1-day toric control (Control) contact lens in the other eye. Patient will wear as an unmatched pair, per predetermined randomization schedule (to determine which eye receives the Test or Control contact lens).
  Interventions: Device: 1-day toric test contact lens; Device: 1-day toric control contact lens
- 1-day toric control contact lens (Active Comparator): Each subject will wear the 1-day toric test (Test) lens in one eye and 1-day toric control (Control) contact lens in the other eye. Patient will wear as an unmatched pair, per predetermined randomization schedule (to determine which eye receives the Test or Control contact lens).
  Interventions: Device: 1-day toric test contact lens; Device: 1-day toric control contact lens

INTERVENTIONS:
Device: 1-day toric test contact lens — somofilcon A 1-day toric test contact lens
  Other Names: Test contact lens; Invigor toric 1-day contact lens
Device: 1-day toric control contact lens — somofilcon A 1-day toric control contact lens
  Other Names: Control contact lens

SUMMARY:
An evaluation of the clinical performance of the 1-day toric test contact lens compared to the 1-day toric control contact lens over one hour of lens wear.

DETAILED DESCRIPTION:
A non-dispensing, double-masked, randomized, contralateral study comparing the 1-day toric test contact lens against the 1-day toric control contact lens to evaluate the clinical performance over one hour of lens wear. Each subject will be randomized to wear the test lens in one eye and the control lens in the other eye for each pair of lenses.

Each subject will be asked to wear four pairs of contact lenses in the study

ELIGIBILITY:
Inclusion Criteria:

* Has had a self-reported oculo-visual examination in the last two years.
* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Is correctable to a visual acuity of 20/40 or better (in each eye) with their habitual vision correction or 20/20 best-corrected.
* Currently wears soft contact lenses.
* Has clear corneas and no active ocular disease.
* Has not worn lenses for at least 12 hours before the examination

Exclusion Criteria:

* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pete S Kollbaum, OD PhD, Principal Investigator — Clinical Optics Research Lab (CORL) Indiana University School of Optometry, Indiana University
Locations (1):
- Clinical Optics Research Lab (CORL) Indiana University School of Optometry, Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Test Contact Lenses / Control Contact Lenses: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye for 1 hour.
  Four different powers of test and control lens were used. There was a 15-minute wash-out period between the two lens pairs
  1-day toric test contact lens 1: Invigor 1-day toric test contact lens -1.00 -1.75 x 180, -1.00 -1.75 x 090, -6.00 -1.75 x 180, -6.00 -1.75 x 090
  1-day toric control contact lens 1: somofilcon A 1-day toric control contact lens -1.00 -1.75 x 180, -1.00 -1.75 x 090, -6.00 -1.75 x 180, -6.00 -1.75 x 090
Period: Pair 1 Test / Control Dispense
Arm/Group | Test Contact Lenses / Control Contact Lenses
Started | 10; 20 Eyes
Completed | 10; 20 Eyes
Not Completed | 0; 0 Eyes
Period: Pair 1 Test /Control Follow up
Arm/Group | Test Contact Lenses / Control Contact Lenses
Started | 10; 20 Eyes
Completed | 10; 20 Eyes
Not Completed | 0; 0 Eyes
Period: Pair 2 Test / Control Dispense
Arm/Group | Test Contact Lenses / Control Contact Lenses
Started | 10; 20 Eyes
Completed | 10; 20 Eyes
Not Completed | 0; 0 Eyes
Period: Pair 2 Test /Control Follow up
Arm/Group | Test Contact Lenses / Control Contact Lenses
Started | 10; 20 Eyes
Completed | 10; 20 Eyes
Not Completed | 0; 0 Eyes
Period: Pair 3 Test / Control Dispense
Arm/Group | Test Contact Lenses / Control Contact Lenses
Started | 10; 20 Eyes
Completed | 10; 20 Eyes
Not Completed | 0; 0 Eyes
Period: Pair 3 Test /Control Follow up
Arm/Group | Test Contact Lenses / Control Contact Lenses
Started | 10; 20 Eyes
Completed | 10; 20 Eyes
Not Completed | 0; 0 Eyes
Period: Pair 4 Test / Control Dispense
Arm/Group | Test Contact Lenses / Control Contact Lenses
Started | 10; 20 Eyes
Completed | 10; 20 Eyes
Not Completed | 0; 0 Eyes
Period: Pair 4 Test /Control Follow up
Arm/Group | Test Contact Lenses / Control Contact Lenses
Started | 10; 20 Eyes
Completed | 10; 20 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Visibility of Toric Mark
Description: Toric Mark visible or not visible. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 1 hour
Population: The primary objective of the study was to validate the clinical performance of test and control contact lenses. The various lens powers and axis of test and control lenses were combined as the primary objective was not to validate different power of test and control lenses.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Contact Lenses
Groups:
- Test Contact Lenses: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used and all the data was combined.
  1-day toric test contact lens: Invigor 1-day toric test contact lens.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
- Control Contact Lenses: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used and all the data was combined.
  1-day toric control contact lens: somofilcon A 1-day toric control contact lens.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact Lenses) | 40 | 40
percentage of participants
  Visible | 100 | 100
  Not Visible | 0 | 0

2. Primary Outcome: Degree of Lens Orientation
Description: Average of lens toric mark mislocation from the resting toric mark away from the 6 o'clock position - measured in degrees.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Contact Lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact Lenses) | 40 | 40
Degrees | 0 (7) | -1 (7)

3. Primary Outcome: Degree of Lens Orientation
Description: as for outcome 2
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Contact Lenses
Groups:
- Control Contact Lenses: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used.
  1-day toric control contact lens: somofilcon A 1-day toric control contact lens.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact Lenses) | 40 | 40
Degrees | 1 (6) | 0 (7)

4. Primary Outcome: Degree of Lens Orientation
Description: as for outcome 2
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Contact lenses
Groups:
- Test Contact Lenses: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used.
  1-day toric test contact lens: Invigor 1-day toric test contact lens. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
Degrees | -1 (6) | -1 (6)

5. Primary Outcome: Toric Stability
Description: Toric stability (maximal and minimal differences between extreme gazes) measured in degrees for up, down, right, and left gazes.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Contact Lenses
Groups:
- Test Contact Lenses: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used.
  1-day toric test contact lens 1: Invigor 1-day toric test contact lens.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact Lenses) | 40 | 40
Degrees | 4 (3) | 4 (3)

6. Primary Outcome: Toric Stability
Description: Rotational stability (maximal and minimal differences between extreme gazes) measured in degrees for up, down, right, and left gazes.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
Degrees | 5 (3) | 4 (3)

7. Primary Outcome: Degree of Rotational Recovery
Description: Rotational Recovery for nasal and temporal - measured in degrees. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (contact lenses) | 40 | 40
Degrees
  Nasal | 16 (9) | 15 (10)
  Temporal | 10 (10) | 10 (9)

8. Primary Outcome: Degree of Rotational Recovery
Description: as for outcome 7
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Contact lenses
Groups:
- Test Contact Lenses: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used.
  1-day toric test contact lens 1: Inigor 1-day toric test contact lens. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
Degrees
  Nasal | 16 (9) | 12 (10)
  Temporal | 9 (10) | 10 (10)

9. Primary Outcome: Toric Fit Acceptance
Description: Toric fit acceptance and preference scale 0-4 (0 = can't be worn, 4 = optimum). Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Contact Lenses
Groups:
- Control Contact Lens: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used.
  1-day toric control contact lens: somofilcon A 1-day toric control contact lens.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Arm/Group | Test Contact Lenses | Control Contact Lens
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact Lenses) | 40 | 40
units on a scale | 3.5 (0.2) | 3.4 (0.2)

10. Primary Outcome: Toric Fit Acceptance
Description: as for outcome 9
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Contact Lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact Lenses) | 40 | 40
units on a scale | 3.5 (0.2) | 3.4 (0.3)

11. Primary Outcome: Toric Fit Preference
Description: Investigator's toric fitting preference - Test lens , No Preference , Control lens.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Contact Lenses
Groups:
- Overall Study: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Arm/Group | Overall Study
Number analyzed (Participants) | 10
Number analyzed (Contact Lenses) | 40
percentage of eyes
  Test Lens | 23
  No Preference | 69
  Control Lens | 8

12. Primary Outcome: Toric Fit Preference
Description: Investigator's toric fitting preference - Test lens, No Preference, Control lens.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 1 hour
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Contact Lenses
Arm/Group | Overall Study
Number analyzed (Participants) | 10
Number analyzed (Contact Lenses) | 40
percentage of eyes
  Test Lens | 33
  No Preference | 57
  Control Lens | 10

13. Secondary Outcome: Measurement of Lens Horizontal Centration
Description: Measurement of Lens Horizontal Centration in millimeters. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 15 Minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: Contact Lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact Lenses) | 40 | 40
millimeters (mm) | -0.08 (0.24) | -0.05 (0.21)

14. Secondary Outcome: Measurement of Lens Horizontal Centration
Description: as for outcome 13
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: Contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
millimeters (mm) | -0.06 (0.22) | -0.08 (0.21)

15. Secondary Outcome: Measurement of Lens Vertical Centration
Description: Lens Horizontal centration measured in mm. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: Contact lenses
Groups:
- Control Contact Lenses: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used. Both lens type and powers were randomized.
  1-day toric control contact lens: somofilcon A 1-day toric control contact lens.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
millimeters (mm) | 0.34 (0.22) | 0.34 (0.21)

16. Secondary Outcome: Measurement of Lens Vertical Centration
Description: Lens Horizontal centration measured in mm. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: Contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
millimeters (mm) | 0.32 (0.19) | 0.27 (0.26)

17. Secondary Outcome: Measurement of Lens Movement
Description: Measurement of lens movement in millimeters. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (contact lenses) | 40 | 40
millimeters (mm) | 0.26 (0.09) | 0.25 (0.08)

18. Secondary Outcome: Measurement of Lens Movement
Description: Measurement of lens movement in millimeters. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: Contact Lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact Lenses) | 40 | 40
millimeters (mm) | 0.25 (0.08) | 0.24 (0.08)

19. Secondary Outcome: Lens Push-Up
Description: Lens push-up measured in percentage. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: Contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
percentage | 45 (6) | 47 (6)

20. Secondary Outcome: Lens Push-Up
Description: Lens push-up measured in percentage. Data for all 4 pairs were combined and analyzed (n=40 control lenses).
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: Contact Lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact Lenses) | 40 | 40
percentage | 47 (5) | 47 (6)

21. Secondary Outcome: Primary Lens Gaze Lag
Description: Primary lens gaze lag measured in millimeters. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: Contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
millimeters (mm) | 0.20 (0.08) | 0.21 (0.08)

22. Secondary Outcome: Primary Lens Gaze Lag
Description: Primary lens gaze lag measured in millimeters. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: Contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
millimeters (mm) | 0.20 (0.06) | 0.19 (0.08)

23. Secondary Outcome: General Lens Fit Acceptance
Description: General lens fit acceptance and preference scale 0-4 (0 = unacceptable, 4 = optimal).
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
units on a scale | 3.4 (0.2) | 3.4 (0.2)

24. Secondary Outcome: General Lens Fit Acceptance
Description: as for outcome 23
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (Contact lenses) | 40 | 40
units on a scale | 3.4 (0.2) | 3.4 (0.2)

25. Secondary Outcome: Up Gaze Lag
Description: Up gaze lag measured in millimeters. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: contact lenses
Arm/Group | Test Contact Lenses | Control Contact Lenses
Number analyzed (Participants) | 10 | 10
Number analyzed (contact lenses) | 40 | 40
millimeters (mm) | 0.25 (0.10) | 0.25 (0.09)

26. Secondary Outcome: Up Gaze Lag
Description: Up gaze lag measured in millimeters. Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: contact lenses
Groups:
- Control Contact Lense: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used.
  1-day toric control contact lens: somofilcon A 1-day toric control contact lens.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Arm/Group | Test Contact Lenses | Control Contact Lense
Number analyzed (Participants) | 10 | 10
Number analyzed (contact lenses) | 40 | 40
millimeters (mm) | 0.22 (0.08) | 0.22 (0.08)

27. Secondary Outcome: General Lens Fit Preference
Description: Investigator's general lens fit preference - Test lens, No preference, Control lens.
  Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Contact lenses
Groups:
- Overall Study: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used.
  1-day toric test contact lens 1: Invigor 1-day toric test contact lens
  1-day toric control contact lens 1: somofilcon A 1-day toric control contact lens Data for all 4 pairs were combined and analyzed (n=40 contact lenses).
Arm/Group | Overall Study
Number analyzed (Participants) | 10
Number analyzed (Contact lenses) | 40
percentage of eyes
  Test Lens | 5
  No preference | 92
  Control lens | 3

28. Secondary Outcome: General Lens Fit Preference
Description: as for outcome 27
Time Frame: 1 hour
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: contact lenses
Arm/Group | Overall Study
Number analyzed (Participants) | 10
Number analyzed (contact lenses) | 40
percentage of eyes
  Test Lens | 3
  No preference | 94
  Control lens | 3

ADVERSE EVENTS:
Time Frame: From dispense up to 1 hour on each pair of lenses.
Groups:
- Test Contact Lenses: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used and the data was combined as the primary objective of the study was to validate the clinical performance of test and control contact lenses. The various lens powers and axis of test and control lenses were combined as the primary objective was not to validate different power of test and control lenses.
  1-day toric test contact lens -1.00 -1.75 x 180, -1.00 -1.75 x 090, -6.00 -1.75 x 180, -6.00 -1.75 x 090
- Control Contact Lenses: Subjects were randomized to wear 1-day toric test lens in one eye and 1-day toric control contact lens in the other eye. Four different powers of test and control contact lenses were used and the data was combined as the primary objective of the study was to validate the clinical performance of test and control contact lenses. The various lens powers and axis of test and control lenses were combined as the primary objective was not to validate different power of test and control lenses.
  1-day toric control contact lens -1.00 -1.75 x 180, -1.00 -1.75 x 090, -6.00 -1.75 x 180, -6.00 -1.75 x 090
Arm/Group | Test Contact Lenses | Control Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT04016623/Prot_SAP_000.pdf